CLINICAL TRIAL: NCT07302217
Title: Effect of Technology-Assisted Intervention Program on Postoperative Handgrip Strength, Muscle Endurance, and Psychological Distress in Patients With Pulmonary Nodules
Brief Title: Effect of Technology-Assisted Preoperative Home Exercise on Postoperative Handgrip Strength, Muscle Endurance, and Psychological Distress in Patients With Pulmonary Nodules Undergoing Video-Assisted Thoracoscopic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202509080RINB
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Nodules
Keywords: exercise; APP LINE; Lung nodule
MeSH Terms: conditions — Multiple Pulmonary Nodules; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study uses a single-group assignment model without a control group. All participants receive the LINE-based preoperative exercise intervention, and outcomes are compared across baseline, pre-surgery, and two-week postoperative assessments.
Masking Description: No masking was implemented because all participants and investigators were aware of the intervention procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Technology-Assisted Preoperative Home-Based Exercise Program (Experimental): Participants in this arm will receive a technology-assisted preoperative home-based exercise program delivered through a LINE APP. The program includes aerobic, resistance, and breathing exercises performed for at least one week before surgery. Educational messages, reminders, and interactive feedback are provided through the LINE platform to support exercise adherence.
  Interventions: Behavioral: Technology-Assisted Preoperative Home-Based Exercise Program

INTERVENTIONS:
Behavioral: Technology-Assisted Preoperative Home-Based Exercise Program — This behavioral intervention uses a technology-assisted approach to deliver preoperative home-based exercise training for patients scheduled to undergo video-assisted lung nodule resection. The intervention integrates a LINE Official Account with an automated LINE Bot that provides exercise instructions, educational materials, reminders, and self-report mechanisms.
  The exercise program is based on published preoperative home-exercise protocols for lung cancer surgery patients. It includes:
  1. Aerobic exercise - walking or marching in place for 30 minutes, three times per week;
  2. Resistance training - six exercises (high-knee marching, bridging, sit-to-stand, shoulder press, biceps curl, heel raise), performed twice weekly (non-consecutive), 30 repetitions each;
  3. Breathing exercises - pursed-lip and diaphragmatic breathing, 10 repetitions each, three times per week;
  4. Warm-up and cool-down for 5 minutes before and after exercise. The LINE Bot system provides video demonstration

SUMMARY:
This study aims to evaluate the effects of a technology-assisted preoperative home-based exercise program, delivered through a LINE Official Account and LINE BOT, on postoperative hand-grip strength, muscle endurance, and psychological distress in patients undergoing thoracoscopic pulmonary nodule resection. The study adopts a single-group pretest post-test design and plans to recruit 60 eligible patients.

The intervention consists of at least one week of home exercise training before surgery, incorporating aerobic, resistance, and breathing exercises. Education, guidance, and interactive feedback are provided through the LINE platform to support adherence and exercise performance. Outcomes will be assessed at three time points: baseline (T0), immediately before surgery (T1), and two weeks after surgery (T2).

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality in Taiwan, and pulmonary nodule resection is a common surgical intervention. Patients often experience postoperative declines in physical function, including hand-grip strength, muscle endurance, and aerobic capacity, along with increased psychological distress such as anxiety and depression. Preoperative rehabilitation has been shown to improve peri-operative outcomes; however, traditional in-person programs are often limited by time constraints, travel burden, and access barriers. Technology-assisted remote health interventions have emerged as a feasible approach to enhancing patient engagement and extending preoperative support.

This study aims to evaluate the effectiveness of a technology-assisted preoperative home-based exercise program delivered through a LINE Official Account and LINE BOT platform. The program is designed to improve postoperative hand-grip strength, muscle endurance, body composition, and psychological distress among patients undergoing thoracoscopic pulmonary nodule resection. The study adopts a quasi-experimental single-group pretest-posttest design and plans to enroll approximately 60 eligible participants.

The intervention includes at least one week of home-based exercise training before surgery and consists of aerobic exercises (such as walking or marching), resistance training movements (including high-knee marching, sit-to-stand, and other functional muscle-strengthening exercises), and breathing exercises (including pursed-lip breathing and diaphragmatic breathing). Educational materials, reminders, guidance, and interactive feedback will be delivered through the LINE platform to enhance adherence, reinforce correct techniques, and support patient engagement.

Outcome assessments will be conducted at three time points: baseline (T0) during the outpatient visit when surgery is scheduled; immediately before surgery at hospital admission (T1); and two weeks after surgery (T2). Primary outcomes include hand-grip strength and muscle endurance, while secondary outcomes include body composition and psychological distress (anxiety and depression).

This study is expected to establish a feasible, sustainable, and flexible model for technology-assisted preoperative health promotion. Findings may provide evidence for integrating digital health tools into peri-operative care pathways to support enhanced recovery following thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pulmonary nodules who are scheduled to undergo video-assisted thoracoscopic surgery for nodule resection (including wedge resection, segmentectomy, or lobectomy).
2. Aged 20 years or older and assessed by a healthcare provider as medically suitable to participate in exercise training.
3. At least one week between the date of enrollment and the scheduled surgery.
4. Willing to provide written informed consent and complete all study procedures, including joining the LINE Official Account, participating in the exercise training, completing questionnaires, and undergoing outcome assessments.

Exclusion Criteria:

1. Metastatic tumors or contraindications to exercise participation.
2. Engagement in regular aerobic or resistance exercise within the past month (defined as ≥2 sessions per week, ≥30 minutes per session).
3. Inability to communicate in Mandarin or Taiwanese.
4. Inability to use technology-assisted applications (e.g., LINE APP).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-17 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hand-grip Strength | Before surgery (T0) to 2 weeks post-surgery (T2)
  Hand-grip strength will be measured using a calibrated handheld dynamometer. Measurements will be collected at three time points:
  Baseline at outpatient visit when surgery is scheduled (T0), Preoperative assessment on the day of admission (T1), Two weeks after surgery (T2). The primary outcome is the change in dominant-hand grip strength from T0 to T2. Higher values indicate greater muscle strength. The measure reflects postoperative functional recovery and the effectiveness of the technology-assisted preoperative exercise program.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The plan for sharing individual participant data (IPD) has not yet been determined. Decisions regarding data sharing will depend on institutional policies, ethical considerations, and data privacy regulations. IPD will only be shared if appropriate safeguards and approvals are in place.